CLINICAL TRIAL: NCT06858020
Title: NoPro - Norwegian Hernia Prophylaxis Study: Onlay Mesh Versus Small Bite Suture Technique Closure of Midline Laparotomies
Brief Title: NoPro - Norwegian Hernia Prophylaxis Study
Acronym: NoPro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 761933
Record Dates: First submitted 2025-02-10; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Incisional Hernia After Midline Laparotomy; Quality of Life (QOL); Burst Abdomen; Surgical Site Infections
Keywords: prophylactic mesh; onlay; incisional hernia; midline laparotomy
MeSH Terms: conditions — Surgical Wound Infection; Incisional Hernia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The radiologists who interpret the CT scans after 12 months evaluating if the patient has developed an incisional hernia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh group (Experimental): The patients in the mesh group are closed with small bites technique and in addition receiving an onlay polypropylene mesh when closing the fascia in midline laparotomies. These patients receive a subcutaneous drain to prevent seroma.
  Interventions: Procedure: Prophylactic polypropylene onlay mesh
- Suture group (No Intervention): The patients in the suture group are closed with small bites technique.

INTERVENTIONS:
Procedure: Prophylactic polypropylene onlay mesh — The patients in the mesh group are closed with small bites technique and in addition receiving an onlay polypropylene mesh when closing the fascia in midline laparotomies.
  Arms: Mesh group

SUMMARY:
A multicenter randomized controlled trial comparing midline laparotomy closures using the small-bite suture technique alone to those using the small-bite suture technique with an additional onlay prophylactic polypropylene mesh. The primary endpoint is the incidence of incisional hernias in both groups after one year.

DETAILED DESCRIPTION:
An incisional hernia (IH) is a defect in the abdominal wall at the site of a surgical scar, leading to the protrusion of abdominal contents through the defect. It is a common complication following midline laparotomy, with incidence rates ranging from 9% to 40% in the general population, and up to 69% in high-risk patients. Several studies have been conducted on the prevention of IH, and one established intervention is the use of a synthetic mesh to reinforce the suture closure of the abdomen after midline laparotomy. However, the use of mesh in this context is not widespread in Norway, and there are no Norwegian studies on IH prevention following midline laparotomy. This study aims to contribute to the broader knowledge base and encourage Norwegian surgeons to consider using prophylactic meshes.

The study will involve three Norwegian hospitals: Hamar Hospital, Gjøvik Hospital, and Lillehammer Hospital. Participants will be patients scheduled for midline laparotomy at these hospitals who consent to participate, meet the inclusion criteria, and do not meet any exclusion criteria. Participants will be randomly assigned to two groups, each receiving a different variation of fascia closure during laparotomy. One group will undergo closure using the standard small-bites technique only, while the other group will undergo closure with the small-bites technique in addition to an onlay polypropylene mesh.

The primary outcome is the occurrence of incisional hernia one year after surgery, identified through clinical examination and CT scan. Additionally, surgical site occurrences (e.g., hematoma, infection, seroma, wound dehiscence) will be recorded four to six weeks post-surgery. Quality of life and pain levels will also be assessed at both four to six weeks and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Surgery predominantly done my midline laparotomy
* Age 18 years old or older
* Written consent by patient/family
* Midline laparotomy with delayed closure
* No exclusion criteria

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Previous abdominal midline hernia mesh repair
* Abdominal compartment syndrome
* Linea alba closure not possible
* Life expectancy under six months
* Hernia in the midline with transverse diameter lager than 2 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia | 12 months
  Incisional hernia occurrence will be evaluated clinically and by CT examination after 12 months

SECONDARY OUTCOMES:
Quality of Life | 4-6 weeks and 1 year
  Quality of life will be measured preoperatively for elective patients and after 4-6 weeks and after 1 year for all patients. Quality of life will be measured using 5-level EQ-5D version (EQ-5D-5L) provided by the EuroQol group. The system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Level of pain | 4-6 weeks and 1 year
  Pain level will be measured preoperatively for elective patients and after 4-6 weeks and after 1 year for all patients. The level will be measured using VAS-scale from 0 to 10 where 0 is explained as "no pain" and 10 is explained as "the worst pain you can possibly imagine".
Symptomatic surgical site occurrence (SSO) | 4-6 weeks
  Symptomatic surgical site occurrence (SSO)when the patient it discharged and after 4-6 weeks. Surgical site occurence including seroma, hematoma, wound dehiscence and infection.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Martin Rekkedal, MD BBA, Study Chair — Chief of surgery Hamar Hospital
Locations (1):
- Innlandet Hospital Trust, Hamar, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT06858020/Prot_000.pdf
  • Informed Consent Form (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT06858020/ICF_001.pdf